CLINICAL TRIAL: NCT06028295
Title: Clinical-instrumental Evaluation of the Efficacy of Two Dietary Supplements Claiming Anti-hair Loss Properties and Hair Strength Improvement. A Double-blind, Randomized, Placebo-controlled Study
Brief Title: Evaluation of the Efficacy of Two Dietary Supplements on Hair Loss and Hair Aspect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT0003622/23
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wheat Polar Lipid Complex Oil (Experimental): Dietary supplement - Wheat Polar Lipid Complex (Oil)
  Interventions: Dietary Supplement: Wheat Polar Lipid Complex Oil
- Wheat Polar Lipid Complex Powder (Experimental): Dietary supplement - Wheat Polar Lipid Complex (Powder)
  Interventions: Dietary Supplement: Wheat Polar Lipid Complex Powder
- Placebo (Placebo Comparator): Dietary supplement - Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wheat Polar Lipid Complex Oil — The study foresees the intake of 2 capsules per day during 84 days
  Arms: Wheat Polar Lipid Complex Oil
Dietary Supplement: Wheat Polar Lipid Complex Powder — The study foresees the intake of 2 capsules per day during 84 days
  Arms: Wheat Polar Lipid Complex Powder
Dietary Supplement: Placebo — The study foresees the intake of 2 capsules per day during 84 days
  Arms: Placebo

SUMMARY:
The study is aimed to assess the efficacy of two dietary supplements composed of a Wheat Polar Lipid Complex (WPLC) in oil or powder form in reducing hair loss and improving hair aspect.

DETAILED DESCRIPTION:
A double blind, parallel groups, placebo-controlled study is carried out on 90 healthy female subjects aged between 18 and 65 years old with all hair type showing diffuse and temporary hair shedding with a proportion of hair in telogen phase >15%. The study foresees 84 days of products intake. Evaluations of the parameters under study are performed at baseline, after 56 and 84 days of products consumption.

ELIGIBILITY:
Inclusion criteria :

* Healthy female subjects,
* Caucasian ethnicity,
* Age between 18 and 65 years old (extremes included),
* All hair type included,
* Subject showing acute hair shedding (duration less than 6 months) due to fatigue, seasonal change, deficiency of vitamins and minerals, stress, change or imbalance of normal daily routing, or emotional stress,
* Women showing a proportion of hair in telogen phase > 15%,
* Subjects complaining brittle and thin hair,
* Subjects who stopped any anti hair loss treatment at least 3 months prior the study,
* Subjects agreeing not to take any treatment (oral or topic) able to interfere with the hair growth, diameter or fall during the whole study duration,
* Subjects who have not been involved in any other similar study in the last 3 months,
* Subjects registered with health social security or health social insurance, Subjects able to understand the language used in the investigation center and the information given
* Subjects able to comply with the protocol and follow protocol's constraints and specific requirements
* Willingness to use the same products for hair care during all the study period
* Willingness not to cut hair for all the study length.
* Subjects having signed their written Informed Consent form (ICF) for their participation in the study and a photograph authorization.

Exclusion Criteria:

* Subject does not meet the inclusion criteria,
* Subject is taking part or planning to participate to another clinical study in the same or in another investigation centre,
* Subject is deprived of freedom by administrative or legal decision or under guardianship,
* Subject is admitted in a sanitary or social facilities,
* Subject is planning an hospitalization during the study,
* Subject has participated in another clinical study with anti-hair loss product or treatment within the last 3 months before the inclusion visit,
* Subject is breastfeeding, pregnant or not willing to take necessary precautions to avoid pregnancy during the study (for the women of childbearing potential),
* Subject has started or changed oestrogen-progesterone contraception or hormonal treatment, within the 3 months prior to the study or foreseeing it for the duration of the study,
* Subject having an acute, chronic or progressive illness liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements,
* Subject is in course of a long-treatment or intending to have one considered by the Investigator liable to interfere with the study data or incompatible with the study requirements,
* Subject having a skin/scalp condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements,
* Subject having personal history of cosmetic, drug, domestic products or food supplements allergy,
* Subject having food disorders,
* Subject who has any other hair disorder or hair disease (female pattern hair loss, any type of alopecia...),
* Subject having excessive and/or fluctuating hair shedding for more than 6 months,
* History or clinical signs of hyperandrogenemia (menstrual cycle >35 days and hirsutism and acne),
* Systemic treatment affecting the hair growth taken for more than 4 consecutive weeks during the last 24 weeks before inclusion visit: retinoids, anti-mitotic, cytotoxic drugs other than antineoplastic, anti-androgens (spironolactone, flutamide), androgens, anti-epileptic agents, interferon alpha,
* Systemic or local androgenetic alopecia treatment or product, taken or applied (Minoxidil, Aminexil, Finasteride, Dutasteride, cosmetic solution or capsules with vitamin B, zinc, caffeine...) for more than 4 consecutive weeks during the last 24 weeks before the inclusion visit,
* Any other topical treatment applied on the scalp (non-steroidal anti-inflammatory, ketoconazole...) within the last 2 weeks before the inclusion visit,
* No hair wash in the 48 hours before each visit,
* Any following hair care within the last 2 weeks before each visit: dandruff shampoo, antifungal shampoo, dyeing, bleaching, perm,
* Any hair care product applied on the scalp between the last shampoo and the inclusion visit (e.g. gel, hairspray, wax, foam...),
* Radiotherapy, chemotherapy at any time,
* Scalp surgery (hair transplants, laser) at any time.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Telogen hair proportion | Baseline
  Phototrichogram
Telogen hair proportion | 56 days
  Phototrichogram
Telogen hair proportion | 84 days
  Phototrichogram

SECONDARY OUTCOMES:
Anagen hair proportion | Baseline
  Phototrichogram
Anagen hair proportion | 56 days
  Phototrichogram
Anagen hair proportion | 84 days
  Phototrichogram
Hair growth | 84 days
  Hair length after shaving
Hair elasticity | Baseline
  Hair elongation using dynamometer
Hair elasticity | 84 days
  Hair elongation using dynamometer
Hair loss | Baseline
  Pull test
Hair loss | 56 days
  Pull test
Hair loss | 84 days
  Pull test
Self-assessment of product efficacy | 84 days
  Questionnaire (20 questions with 4 possible answers : completely agree / agree / disagree / completely disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Ileana De Ponti, Study Director — Complife Italia S.r.l
Locations (1):
- Complife Italia srl, Milan, Italy